# MEDICA LA POSITION DE

#### MEDICAL UNIVERSITY OF WARSAW

Department of Neurosurgery Head: Professor Andrzej Marchel, MD, PhD

Prophylactic Use of Dural Tenting Sutures in Elective Craniotomies – Is It Necessary? A multicenter Randomised Study.

STUDY PROTOCOL

14/01/2020

### 1. Study Identification

Unique Protocol identification Number:

KB/106/2018

Brief Title:

Dural tenting sutures in neurosurgery - is it necessary?

Official Title:

Prophylactic use of dural tenting sutures in elective craniotomies - is it necessary? A multicentre randomised study.

Acronym:

Study Type:
Interventional

#### 2. STUDY STATUS

Record Verification Date:

June 2018

Overall Recruitment Status:

Recruiting

Study Start Date:

September 7, 2018

Primary Completion Date:

Anticipated September 1, 2021

Study Completion Date:

Anticipated April 1, 2022

#### 3. SPONSOR/COLLABORATORS

Responsible Party, by Official Title:

Sponsor

Investigator Information:

Investigator Name:

Przemysław Kunert

Investigator Official Title:

MD, PhD, Vice Chair of Department of Neurosurgery
Investigator Affiliation:

Department of Neurosurgery, Medical University of Warsaw
Investigator Information:
Investigator Name:
Łukasz Przepiórka
Investigator Official Title:

Investigator Affiliation:
Department of Neurosurgery, Medical University of Warsaw

Name of the Sponsor:
Medical University of Warsaw

#### 4. OVERSIGHT

Studies a U.S. FDA-regulated Drug Product: Studies a U.S. FDA-regulated Device Product: No Device Product Not Approved or Cleared by U.S. FDA: No Post Prior US FDA Approval or Clearance: Investigational New Drug Application(IND)/Investigational Device Exemption (IDE) Information: U.S. Food and Drug Administration IND or IDE: No Human Subjects Review: Human Subjects Protection Review Board Status: Submitted, approved Board Approval Number: KB / 106 / 2018 Board Name: Komisja Bioetyczna przy Warszawskim Uniwersytecie Medycznym (Bioetics Comitee, Medical University of Warsaw)

Medical University of Warsaw

Board Contact:

Phone:
+48 22 57 20 30

Email:

komisja.bioetyczna@wum.edu.pl

Address:
ul. Żwirki I Wigury nr 61, 02-091 Warszawa

Data Monitoring Committee:

Yes

FDA Regulated Intervention:

No

Section 801 Clinical Trial:

#### 5. STUDY DESCRIPTION

Brief Summary (using lay language:)

This study evaluates the necessity of dural tenting sutures in craniotomies. The sutures elevate the dura, a layer between the brain and skull. Supposedly, by doing so, they prevent blood collecting between dura mater and the skull. These blood collections, called epidural hematomas, contributed greatly to postoperative mortality in the early days of neurosurgery. There have been several reports questioning the ongoing need for them in neurosurgery, thanks to modern hemostatic techniques. Moreover, it has been published in the literature, and is a common knowledge as well, that some neurosurgeons do not use these sutures at all, and do not have worse outcomes than their colleagues.

In this study, half of the randomly assigned participants will undergo craniotomy without dural tenting sutures and will be considered an intervention group. The other half will undergo craniotomy with these sutures.

Detailed Description:

In the early days of neurosurgery, epidural hemorrhages (EDH) contributed to a high mortality rate after craniotomies. Almost a century ago Walter Dandy reported dural tenting sutures as an effective way of preventing postoperative EDH. Over time, his technique gained in popularity and significance to finally become a neurosurgical standard.

Yet, there have been several retrospective reports questioning the ongoing need for dural tenting sutures. Dandy's explanation that the hemostasis under hypotensive conditions is deceiving and eventually causes EDH may be obsolete. These days, proper intra- and postoperative care, including maintenance of normovolemia and normotension and the use of modern hemostatic agents, may be enough for effective hemostasis. Evading of this suturing technique by some surgeons supports this argument even further.

Thus, there is a fundamental need to evaluate the necessity of dural tenting sutures in an unbiased, evidence-based manner.

#### 6. CONDITIONS AND KEYWORDS

Primary Disease or Condition Being Studied in the Trial, or the Focus of the Study:

1. Epidural Hematoma

Keywords:

- 1. Craniotomy
- 2. Dural Tenting Suture
- 3. Epidural Hematoma

### 7. STUDY DESIGN (INTERVENTIONAL)

| Primary purpose: |
|---|
| Prevention |
| Study Phase: |
| N/A |
| Interventional Study Model: |
| Parallel |
| Model Description: |
| We plan to include 2000 subjects in this study. Each subject will undergo a craniotomy for unrelated pathology. Each of the subjects will be assigned in random order to an intervention or control group. The intervention group will not have dural tenting sutures during closure of their craniotomy while the control group will have at least three. |
| Both groups will be followed radiologically and clinically, in the exact same manner. |
| Number of Arms: |
| 2 |
| Masking Roles, if Masking: |
| Participant |
| Investigator |
| Outcomes Assessor |
| Masking Description: |
| Due to the nature of the surgical procedures, the surgeon and the rest of the OR medical team will be aware of the current subject's allocation. However, in each case, the specific OR team aware of the subject's allocation will be different from the investigators performing further evaluation of the given subject. The following study procedures will be in place to ensure double-blind administration of the study. |
| Access to the randomization code will be strictly controlled. |
| The surgeon will receive information on subject's allocation after commencing the |

The study blind will be broken:

surgery.

1. During interim monitoring, after recruiting the first 100 patients.

| 2. | On completion of the clinical study and after the study database has been locked. |
|---|---|
| 3. | When patients' safety requires access to allocation data. |
| Allocatio | on: |
| Random | ized |
| Enrollme | nt Type: |
| Anticipa | ted |
| Number | of Participants: |
| 2 000 | |

# 8. ARMS, GROUPS, AND INTERVENTIONS

| | Arm 1: |
|-----------------------------------|--------|
| Arm Type: | |
| No intervention | |
| Arm Title: | |
| No dural tenting sutures | |
| Arm Description: | |
| No dural tenting technique | s |
| | Arm 2: |
| Arm Type: | |
| Active Comparator | |
| Arm Title: | |
| Arm Title: Dural tenting sutures | |

| Intervention 1: |
|-----------------------------|
| Intervention Type: |
| Procedure/Surgery |
| Intervention Name |
| No dural tenting techniques |
| Other Intervention Name 1: |
| No tack-up sutures |
| Other Intervention Name 2: |
| No hitch-up stitches |

| Intervention Description: |
|---|
| Intervention Description: |
| Not applying dural tenting sutures during closure of a craniotomy |
| Intervention 2: |
| Intervention Type: |
| Procedure/Surgery |
| Intervention Name |
| Dural tenting techniques |
| Other Intervention Name 1: |
| No tack-up sutures |
| Other Intervention Name 2: |
| No hitch-up stitches |
| Intervention Description: |
| Applying at least 3 dural tenting sutures during closure of a craniotomy in a usual way |

#### Arm/Interventional Cross-Reference

| | No dural tenting techniques | Dural tenting techniques |
|---|---|---|
| Experimental, no dural tenting sutures | | |
| Active comparator, dural tenting sutures | | |

## 9. OUTCOME MEASURES

| | Outcome 1: |
|---|---|
| F | Primary Outcome Measure: |
| Т | Title: |
| F | Reoperation due to epidural hematoma |
| E | Description: |
| F | Percentage |
| Т | Fime Frame: |
| | During hospitalization for the surgery, approximately 2 days postoperatively |
| | Outcome 2: |
| S | Secondary Outcome Measure: |
| Т | Title: |
| F | Postoperative 30-day mortality |
| E | Description: |
| F | Percentage |
| Т | Time Frame: |
| 3 | 30-day postoperatively |

| Outcome 3: |
|---|
| Secondary Outcome Measure: |
| Title: |
| Postoperative 30-day readmission to a neurosurgical or neurological department |
| Description: |
| Percentage |
| Time Frame: |
| 30-day postoperatively |
| Outcome 4: |
| Secondary Outcome Measure: |
| Title: |
| New neurologic deficit or deterioration of a previous one |
| Description: |
| Specific description of a neurologic deficit |
| Time Frame: |
| During hospitalization, during hospitalisation, as evaluated 5–7 days postoperatively, or earlier if the patient is discharged before the fifth postsurgical day. |
| Outcome 5: |
| Outcome 5: Secondary Outcome Measure: |
| Secondary Outcome Measure: |
| Secondary Outcome Measure: Title: |
| Secondary Outcome Measure: Title: Cerebrospinal fluid leak requiring treatment |
| Secondary Outcome Measure: Title: Cerebrospinal fluid leak requiring treatment Description: |
| Secondary Outcome Measure: Title: Cerebrospinal fluid leak requiring treatment Description: Percentage |
| Secondary Outcome Measure: Title: Cerebrospinal fluid leak requiring treatment Description: Percentage Time Frame: During hospitalization, during hospitalisation, as evaluated 5–7 days postoperatively, or earlier if |
| Secondary Outcome Measure: Title: Cerebrospinal fluid leak requiring treatment Description: Percentage Time Frame: During hospitalization, during hospitalisation, as evaluated 5–7 days postoperatively, or earlier if the patient is discharged before the fifth postsurgical day. |
| Secondary Outcome Measure: Title: Cerebrospinal fluid leak requiring treatment Description: Percentage Time Frame: During hospitalization, during hospitalisation, as evaluated 5–7 days postoperatively, or earlier if the patient is discharged before the fifth postsurgical day. Outcome 6: |
| Secondary Outcome Measure: Title: Cerebrospinal fluid leak requiring treatment Description: Percentage Time Frame: During hospitalization, during hospitalisation, as evaluated 5–7 days postoperatively, or earlier if the patient is discharged before the fifth postsurgical day. Outcome 6: Secondary Outcome Measure: |
| Secondary Outcome Measure: Title: Cerebrospinal fluid leak requiring treatment Description: Percentage Time Frame: During hospitalization, during hospitalisation, as evaluated 5–7 days postoperatively, or earlier if the patient is discharged before the fifth postsurgical day. Outcome 6: Secondary Outcome Measure: Title: |
| Secondary Outcome Measure: Title: Cerebrospinal fluid leak requiring treatment Description: Percentage Time Frame: During hospitalization, during hospitalisation, as evaluated 5–7 days postoperatively, or earlier if the patient is discharged before the fifth postsurgical day. Outcome 6: Secondary Outcome Measure: Title: Deterioration of postoperative headaches over 5 in Numerical Rating Scale |

During hospitalization, during hospitalisation, as evaluated 5–7 days postoperatively, or earlier if

| the patient is discharged before the fifth postsurgical day. |
|---|
| Outcome 7: |
| Secondary Outcome Measure: |
| Title: |
| Epidural collection thickness over 3 mm measured radiographically |
| Description: |
| The thickness of the epidural collection measured in a postoperative CT scan |
| Time Frame: |
| During hospitalization, approximately 1-3 days postoperatively |
| Outcome 8: |
| Secondary Outcome Measure: |
| Title: |
| Midline shift over 5 mm |
| Description: |
| Midline shift caused by the epidural collection measured in a postoperative CT scan |
| Time Frame: |
| During hospitalization, approximately 1-3 days postoperatively |

# 10. ELIGIBILITY

| Sex/Gender: |
|-----------------------------|
| Sex: |
| All |
| Gender-Based: |
| No |
| Age Limits: |
| Minimum Age: |
| 18 |
| Unit of Time: |
| Years |
| Maximum Age: |
| 75 |
| Unit of Time: |
| Years |
| Accepts Healthy Volunteers: |
| No |
| Eligibility Criteria: |

#### Inclusion Criteria:

- Male or female over 18 an under 75 years old
- Qualified for an elective supratentorial craniotomy with a diameter of at least 3 cm
- Glasgow Coma Scale 15 preoperatively
- Modified Rankin Scale 0, 1 or 2 preoperatively

#### Exclusion Criteria:

- Coagulation abnormalities before the surgery
- Revision craniotomy
- Skull base surgery

# 11. CONTACTS, LOCATIONS, AND INVESTIGATOR INFORMATION

| | Central Contact Person: |
|------------------------------|-------------------------|
| First Name: | |
| Przemysław | |
| Last Name or Official Title: | |
| Kunert | |
| Degree: | |
| MD, PhD | |
| Phone: | |
| +48 22 599 25 29 | |
| Email: | |
| przemyslaw.kunert@wum.edu.pl | |
| | Central Contact Backup: |
| First Name: | |
| Łukasz | |
| Last Name or Official Title: | |
| Przepiórka | |
| Degree: | |
| Phone: | |
| +48 22 599 25 75 | |
| Email: | |
| przepiorka@mp.pl | |

| | Overall Study Official 1: |
|-------|--------------------------------------------------------|
| First | t Name: |
| Łuk | casz |
| Las | t Name or Official Title: |
| Prze | epiórka |
| De | gree: |
| Org | ganization/Affiliation: |
| De | partment of Neurosurgery, Medical University of Warsaw |
| Off | icial's Role: |
| stud | dy principal investigator |
| | Overall Study Official 2: |
| First | t Name: |
| Prze | emysław |
| Las | t Name or Official Title: |
| Kur | nert |
| De | gree: |
| MD | , PhD |
| Org | ganization/Affiliation: |
| De | partment of Neurosurgery, Medical University of Warsaw |
| Off | icial's Role: |
| stud | dy principal investigator |
| | Facility Information: |
| Fac | cility Name: |
| Del | partment of Neurosurgery, Medical University of Warsaw |
| City | y: |
| Wa | rsaw |
| Sta | te/Province: |
| Ma | zovian |
| ZIP) | Postal Code: |
| 02- | 097 |
| Со | untry: |
| | and |

| Facility contact: |
|------------------------------|
| First Name: |
| Łukasz |
| Last Name or Official Title: |
| Przepiórka |
| Degree: |
| Phone: |
| +48 22 599 25 75 |
| Email: |
| przepiorka@mp.pl |
| Facility Contact Backup: |
| First name: |
| Przemysław |
| Last Name: |
| Kunert |
| Degree: |
| MD, PhD |
| Phone: |
| +48 22 599 25 29 |
| Email: |
| przemyslaw.kunert@wum.edu.pl |

| Facility Information |
|---|
| Facility Name: |
| Department of Neurosurgery and Oncology of Central Nervous System, Barlicki University Hospital, Medical University of Lodz |
| City: |
| Łódź |
| State/Province: |
| Łódzkie |
| ZIP/Postal Code: |
| 90-153 |
| Country: |
| Poland |
| Individual Site Status: |

| Recruiting |
|------------------------------|
| Facility contact: |
| First Name: |
| Dariusz |
| Last Name or Official Title: |
| Jaskólski |
| Degree: |
| MD, PhD |
| Phone: |
| +48 42 677 67 82 |
| Email: |
| Facility Contact Backup: |
| First name: |
| Last Name: |
| Degree: |
| Phone: |
| Email: |

| Facility Information: |
|---|
| Facility Name: |
| Department of Neurosurgery, Medical University of Silesia, Regional Hospital, Sosnowiec |
| City: |
| Sosnowiec |
| State/Province; |
| Śląskie |
| ZIP/Postal Code; |
| 41-200 |
| Country: |
| Poland |

| In all data of City Charters |
|------------------------------|
| Individual Site Status: |
| Recruiting |
| Facility contact: |
| First Name: |
| Piotr |
| Last Name or Official Title: |
| Ładziński |
| Degree: |
| MD, PhD |
| Phone: |
| +48 32 368 25 51 |
| Email: |
| Facility Contact Backup: |
| First name: |
| Last Name: |
| Degree: |
| Phone: |
| Email: |

| Facility Information: |
|---|
| Facility Name: |
| Neurosurgery and Pediatric Neurosurgery Department in Lublin, Medical University of Lublin, Lublin, Poland |
| City: |
| Lublin |
| State/Province: |
| Lubelskie |

| ZIP/Postal Code: |
|------------------------------|
| 20-954 |
| Country: |
| Poland |
| Individual Site Status: |
| Recruiting |
| Facility contact: |
| First Name: |
| Radosław |
| Last Name or Official Title: |
| Rola |
| Degree: |
| MD, PhD |
| Phone: |
| +48 81 724 41 76 |
| Email: |
| Facility Contact Backup: |
| First name: |
| Dariusz |
| Last Name: |
| Szczepanek |
| Degree: |
| MD, PhD |
| Phone: |
| Email: |

| Facility Information: |
|---|
| Facility Name: |
| Department of Neurosurgery, 10th Military Research Hospital and Polyclinic, Bydgosz, Poland |
| City: |
| Bydgoszcz |
| State/Province: |

| Kuyavian-pomeranian |
|----------------------------------|
| ZIP/Postal Code: |
| 85-681 |
| Country: |
| Poland |
| Individual Site Status: |
| Recruiting |
| Facility contact: |
| First Name: |
| Kamil |
| Last Name or Official Title: |
| Krystkiewicz |
| Degree: |
| MD |
| Phone: |
| +48 261 417 093 |
| Email: |
| Facility Principal Investigator: |
| First name: |
| Marek |
| Last Name: |
| Harat |
| Degree: |
| MD, PhD |
| Phone: |
| Email: |

Facility Information:

Facility Name:

Department of Neurosurgery and Pediatric Neurosurgery, Pomeranian Medical University, Szczecin, Poland

| City: |
|----------------------------------|
| Szczecin |
| State/Province: |
| West Pomeranian |
| ZIP/Postal Code: |
| 71-252 |
| Country: |
| Poland |
| Individual Site Status: |
| Recruiting |
| Facility contact: |
| First Name: |
| Leszek |
| Last Name or Official Title: |
| Sagan |
| Degree: |
| MD, PhD |
| Phone: |
| +48 91 425 35 61 |
| Email: |
| Facility Principal Investigator: |
| First name: |
| Leszek |
| Last Name: |
| Sagan |
| Degree: |
| MD, PhD |
| Phone: |
| Email: |

### 12. IPD SHARING STATEMENT

| Plan to | Share IPD: |
|---------|------------------------------------|
| No | |
| IPD Sha | aring Plan Description |
| IPD Sha | aring Supporting Information Type: |
| IPD Sha | aring Time Frame: |
| IPD Sha | aring Access Criteria: |
| IPD Sha | aring URL: |

#### 13. REFERENCES

| | Citations |
|---|---|
| PubMed Identifier: | |
| 12617233 | |
| Citation | |
| Swayne OB, Horner BM, D<br>Neurosurg. 2002 Dec;16(6 | orward NL. The hitch stitch: an obsolete neurosurgical technique? Br J<br>5):541-4; discussion 544. |
| Results Reference: | |
| No | |
| PubMed Identifier: | |
| 10433304 | |
| Citation | |
| Winston KR. Efficacy of du | ral tenting sutures. J Neurosurg. 1999 Aug;91(2):180-4. |
| Results Reference: | |
| No | |
| PubMed Identifier: | |
| PubMed Identifier: 9732254 | |

| Winston KR. Dural fenting sutures in pediatric neurosurgery. Pediatr Neurosurg. 1998 May;28(5):230-5. |
|---|
| Results Reference: |
| No |
| PubMed Identifier: |
| 12617233 |
| Citation |
| Swayne OB, Horner BM, Dorward NL. The hitch stitch: an obsolete neurosurgical technique? Br J Neurosurg. 2002 Dec;16(6):541-4; discussion 544. |
| Results Reference: |
| No |
| PubMed Identifier: |
| Citation |
| Wadanamby, S. et al., (2016). Is dural hitching necessary to prevent post-operative extradural haemorrhage in craniotomies and craniectomies. Sri Lanka Journal of Surgery. 34(2), pp.11-17. DOI: http://doi.org/10.4038/sljs.v34i2.8262 |
| Results Reference: |
| No |
| Links |
| URL: |
| Description: |
| Available IPD and Supporting Information: |
| Available IPD/Information Type: |
| Available IPD/Information URL: |
| Available ii Djiiiloittaliott akt. |
| Available IPD/Information Identifier: |
| Available IPD/Information Comments: |